CLINICAL TRIAL: NCT00712699
Title: Placebo vs. Extended Release Stimulant Crossover Trial in Preschoolers With ADHD
Brief Title: Effectiveness of an Extended Release Stimulant Medication in Treating Preschool Children With ADHD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baystate Medical Center (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, john fanton, Primary Investigator, Baystate Medical Center
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: F32MH078388 (NIH); F32MH078388 (NIH); DDTR BK-TKFND
Record Dates: First submitted 2008-07-08; First posted 2008-07-10 (Estimated); Last update posted 2013-08-23 (Estimated); Status verified 2013-08

CONDITIONS: Attention Deficit Disorder With Hyperactivity
Keywords: Preschool; Children; ADHD; Medication; Controlled Study; Placebo; Mixed Amphetamine Salts
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — SLI381

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sequence 1: XR-MAS then placebo (Experimental): Depending on whether 1) child has had previous medication trial or 2) is on psychotropic medication at time of screening, children will either enter the washout period of 3 days before extended release mixed amphetamine salts (XR-MAS) or placebo (PBO) is initiated or proceed directly to the active treatment sequence they were randomized to. Participants randomized to Sequence 1 first receive treatment with XR-MAR for 3 weeks and then placebo for 3 weeks. Flexible, forced dosing will start at 5 mg/day for the first week, increase to 10 mg/day for the second week and continue to 15 mg/day on the third week. No washout period otherwise occurs (XR-MAS is not clinically suspected to have lingering effects beyond initial dosing/day of administration), including the crossover week to PBO.
  Interventions: Drug: Sequence 1: XR-MAS then placebo; Drug: Sequence 2 Placebo then XR-MAS
- Sequence 2 Placebo then XR-MAS (Experimental): Depending on whether 1) child has had previous medication trial or 2) is on psychotropic medication at time of screening, children will either enter the washout period of 3 days before extended release mixed amphetamine salts (XR-MAS) or placebo (PBO) is initiated or proceed directly to the active treatment sequence they were randomized to. Participants randomized to Sequence 2 will first receive treatment with PBO for 3 weeks and then XR-MAS for 3 weeks. Flexible, forced dosing will start at 5 mg/day for the first week, increase to 10 mg/day for the second week and continue to 15 mg/day on the third week. No washout period (stimulants are not clinically suspected to have lingering effects beyond initial dosing/day of administration)otherwise occurs, including the crossover week to XR-MAS.
  Interventions: Drug: Sequence 1: XR-MAS then placebo; Drug: Sequence 2 Placebo then XR-MAS

INTERVENTIONS:
Drug: Sequence 1: XR-MAS then placebo — XR-MAS given in non-identifying 5 mg capsules with instructions to start 1 capsule (5 mg/d) for one week, then increase to 2 capsules (10 mg/d) for week two, and 3 caps (15 mg/d) for week 3 following flexible, forced titration based on response and tolerance.
  Other Names: Adderall XR; IND# 58,037
Drug: Sequence 2 Placebo then XR-MAS — PBO given in non-identifying 5 mg capsules with instructions to start 1 capsule (5 mg/d) for one week, then increase to 2 capsules (10 mg/d) for week two, and 3 caps (15 mg/d) for week 3 following flexible, forced titration based on response and tolerance.

SUMMARY:
This study will evaluate the safety and effectiveness of extended release mixed amphetamine salts in treating preschool children with attention deficit hyperactivity disorder.

DETAILED DESCRIPTION:
Attention deficit hyperactivity disorder (ADHD) is a common developmental disorder that affects between 4% and 12% of school-aged children. Children with ADHD often show symptoms of hyperactivity, inattention, inability to sit still, trouble listening, excessive talking, and aggression. ADHD is generally not diagnosed and treated in children less than 6 years old because some symptoms of ADHD are difficult to distinguish from normal behaviors of preschool-aged children. However, some preschool children who exhibit symptoms indicative of ADHD and who have been carefully diagnosed by a health professional may benefit from early treatment to lower risk for functional impairment later in childhood. Currently, environmental changes, parent effectiveness training, and behavior therapy are the commonly used treatments for preschoolers with ADHD symptoms, but not all preschoolers respond well to such behavioral interventions. These children may benefit from medication treatment; however, the safety and effectiveness of ADHD medications in treating preschool-aged children is not well known. Extended release mixed amphetamine salts (XR-MAS), a stimulant medication, is a commonly prescribed and approved medication for treating ADHD in children 6 years and older. Further study is needed to determine how XR-MAS affects preschool-aged children with ADHD symptoms. This study will compare the safety and effectiveness of XR-MAS versus placebo in treating preschool children with ADHD.

Participation in this study will last 6 weeks. All participants will first undergo rigorous psychiatric assessments to confirm their diagnosis of ADHD. Eligible participants will then be assigned randomly to receive treatment with either XR-MAS then placebo or placebo then XR-MAS. Participants will take their assigned XR-MAS or placebo medications for 3 weeks and then cross over to the other medication for an additional 3 weeks of treatment. Rating scale scores will be collected weekly from parents and teachers to assess symptom response and measures of safety.

ELIGIBILITY:
Inclusion Criteria:

* Living at home for at least 6 months with parent or caregiver
* Enrolled in a structured school setting at least 2 half days a week with a minimum of 7 peers
* Full Scale Intelligence Quotient (FSIQ) of 70 or greater OR 72 or greater if bilingual
* Best estimate diagnosis based on clinical interview, Diagnostic Interview Schedule for Children, Child Behavior Checklist, and rating scales scores
* Symptoms present for at least 9 months
* Meets severity criteria for Clinical Global Impression-Severity with score of greater than or equal to 4 and Clinical Global Assessment Scale score of greater than or equal to 55
* Parent/caregiver can commit to 6 weekly sessions, including initial screening exams
* If on current psychotropic medication, will undergo a washout period of at least 3 days before study entry
* Not currently receiving psychotherapy or started psychotherapy within 30 days of study entry

Exclusion Criteria:

* Previous nonresponse to mixed amphetamine salts (defined as 2 weeks of persistent symptoms in spite of doses greater than or equal to 15 mg per day)
* Diagnosis of language-based or cognitive delay of more than 2 standard deviations below same-aged peers or diagnosis of mental retardation
* Pervasive developmental disorder or autism
* Significant developmental disorder (e.g., blindness, deafness, cerebral palsy, epilepsy, psychosis)
* Taking another psychotropic medication that cannot be discontinued
* Serious psychiatric disorder (e.g., bipolar, suicidality, tic disorder)
* Actively taking medication for certain medical conditions (e.g., hypertension, structural cardiac condition, glaucoma, hyperthyroidism)
* Allergy to mixed amphetamine salts
* History of physical, sexual, or emotional abuse that is clinically significant

Ages: 36 Months to 66 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 27 (Actual)
Dates: Start 2008-06; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Composite Parent and Teacher Conners Rating Scale Score | Measured weekly for 6 weeks
Tolerance of extended release mixed amphetamine salts | Measured weekly for 6 weeks

SECONDARY OUTCOMES:
Clinical Global Impression- Improvement Score | Measured weekly for 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: John H. Fanton, MD, Principal Investigator — Baystate Medical Center